CLINICAL TRIAL: NCT00437125
Title: An Open Label Pilot Study on the Tolerability of Duloxetine in the Treatment of Depressed Patients With Parkinson's Disease
Brief Title: Study on the Tolerability of Duloxetine in Depressed Patients With Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11127; F1J-IT-HMFQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Results first posted 2010-08-16 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Major Depressive Disorder; Idiopathic Parkinson Disease
MeSH Terms: conditions — Depressive Disorder, Major; Parkinson Disease | interventions — Duloxetine Hydrochloride

ARMS (1):
- Duloxetine (Experimental): Participants received duloxetine 30 milligram (mg) orally once daily (QD) for 1 week, followed by duloxetine 60 mg orally QD for 11 weeks
  Interventions: Drug: Duloxetine hydrochloride

INTERVENTIONS:
Drug: Duloxetine hydrochloride — Duloxetine 30 milligram (mg) once daily (QD) orally (PO) for 1 week, then duloxetine 60 mg QD PO for 11 weeks
  Other Names: LY248686; Cymbalta

SUMMARY:
This study aims to assess the tolerability of duloxetine, 60mg once daily, in open label fashion, in depressed patients with Parkinson's disease during 12 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Are outpatients, male or female, 30 through 75 years of age
* Meet diagnostic criteria for major depression episode and a clinical diagnosis of idiopathic Parkinson's disease
* Have a clinician-rated 17-item Hamilton Depression Rating Scale (HAMD17) total score greater than or equal to 15, a Beck Depression Inventory (BDI) total score greater than or equal to 13 and a Clinical Global Impression of Severity (CGI-S) score greater than or equal to 3 at both Visit 1 and Visit 2
* Have satisfactory cognitive function
* Have been held on stable dosage of antiparkinsonian medications for at least 4 weeks immediately prior to Visit 1

Exclusion Criteria:

* Any current primary psychiatric diagnosis other than Major depressive episode, and any personality disorder that could interfere with the compliance with the study protocol
* Atypical or secondary parkinsonism due to drugs or diseases with features of Parkinson's disease
* Motor conditions for which it is to be expected to change the antiparkinsonian treatment during the course of the study
* Clinically significant laboratory abnormalities or serious, unstable medical illness
* Lack of response of current episode to two or more adequate courses of antidepressant therapy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- Italy (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ancona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brescia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lido di Camaiore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Messina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pozzilli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 167 participants were screened and 16 participants were screen failures
Period: Overall Study
Arm/Group | Duloxetine
Started | 151
Completed | 119
Not Completed | 32
Not completed — Adverse Event | 12
Not completed — Death | 1
Not completed — Clinical Relapse | 1
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 13
Not completed — Withdrawal by Caregiver | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Duloxetine
Number analyzed (Participants) | 151
Age Continuous [Mean (Standard Deviation); unit: years] | 63.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 66
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 151
Region of Enrollment [Number; unit: participants]
  Italy | 151
Current alcohol consumption by participants [Number; unit: participants]
  no | 130
  yes | 21
Current use of tobacco products by participants [Number; unit: participants]
  no | 140
  yes | 11
Depression in a distant relative of the participant [Number; unit: participants]
  no | 120
  yes | 1
  unknown | 30
Depression in a second degree relative of the participant [Number; unit: participants]
  no | 126
  yes | 25
Depression in mother or father of participant [Number; unit: participants]
  no | 149
  yes | 1
  unknown | 1
Depression in sibling or child of participant [Number; unit: participants]
  no | 150
  yes | 1
Disease stage of the modified Hoen and Yahr staging scale [Number; unit: participants] — Stage 1: unilateral disease; stage 1.5: unilateral plus axial involvement; Stage 2: bilateral disease, without impairment of balance; Stage 2.5: mild bilateral disease with recovery on pull test; Stage 3: mild to moderate bilateral disease, some postural instability, physically independent; Stage 4: severe disability, still able to walk or stand unassisted; Stage 5: wheelchair or bedridden unless aided.
  participants
    unilateral disease | 23
    unilateral plus axial involvement | 16
    bilateral disease, without impairment of balance | 63
    mild bilateral disease | 40
    mild to moderate bilateral disease | 9
Other Axis 1 disorder in distant relative of participant [Number; unit: participants] — Any axis 1 disorder except depressive disorder.
  participants
    no | 119
    yes | 32
Other Axis 1 disorder in parents of participant [Number; unit: participants] — Any axis 1 disorder except depressive disorder.
  participants
    no | 149
    yes | 1
    unknown | 1
Other Axis 1 disorder in second degree relative of participant [Number; unit: participants] — Any axis 1 disorder except depressive disorder.
  participants
    no | 127
    yes | 24
Other Axis 1 disorder in sibling or child of participant [Number; unit: participants] — Any axis 1 disorder except depressive disorder.
  participants
    no | 150
    yes | 1
Presence of major depressive episode diagnosed with Mini International Neuropsychiatric Interview [Number; unit: participants] — The Mini International Neuropsychiatric Interview (MINI) is a standardized diagnostic interview based on Diagnostic and Statistical Manual of Mental Disorders version 4 (DSM-IV) criteria. It was developed as a more concise and easily administered alternative to the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID).
  participants
    no | 2
    yes | 149
Mini Mental State Examination (MMSE) Total Score [Mean (Standard Deviation); unit: units on a scale] — The MMSE is used to screen cognitive functioning and provides measures of orientation, registration (immediate memory), memory, and language functioning. The score range is 0-30; normal: 25-30; mild impairment: 21-24; moderate impairment: 10-20; severe impairment: <10.
  units on a scale | 28.3 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Serious Adverse Events or Other Adverse Events Leading Either to Discontinuation or to Death
Description: The results reported are the number of participants who discontinued the study as a result of an adverse event (serious or other) or death.
Time Frame: baseline through 12 weeks
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 151
participants | 13
Statistical Analysis 1: Comparison: Duloxetine; Test type: Superiority or Other; Percentage = 8.6, 95% CI 1-sided [upper limit 13.3]

2. Secondary Outcome: Change From Baseline to 12 Weeks on the Unified Parkinson's Disease Rating Scale (UPDRS) Total Score
Description: Rating tool to follow the longitudinal course of Parkinson's Disease. It is composed of Section I: Mentation, Behavior, and Mood; Section II: Activities of Daily Living; Section III: Motor Examination; Section IV: Complications of therapy. These are evaluated by interview. Some sections require that multiple grades be assigned to each extremity. Only Sections II and III were rated in this study. A total of 160 points are possible (52 in Section II and 108 in Section III), where 0 represents no disability and 160 indicates maximal grade of disability.
Time Frame: baseline, 12 weeks
Population: All treated participants were included in the analysis population. Last observation carried forward analysis. Two participants were excluded from calculation of change as they had no post-baseline measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 151
units on a scale
  baseline; n=151 | 32.0 (12.6)
  change; n=149 | -0.3 (6.1)
Statistical Analysis 1: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change on the total UDPRS score from baseline to 12-week endpoint; Test type: Superiority or Other; p = 0.5553, t-test, 2 sided — p-value is for total UDPRS score - change. A priori threshold for p-values was 0.05

3. Secondary Outcome: Change From Baseline to 12 Weeks on the UKU (Udvalg for Kliniske Undersogelser: Committee for Clinical Investigations) Side Effect Rating Scale
Description: Clinician-rated scale, providing side effect ratings of psychopharmacological medications. 48 items, each item is rated on a 4-point scale (0=not present; 1=mild; 2=moderate; 3=severe). The test is divided in 6 subscales, total scores for each subscale are calculated based on a weighted secondary scoring system. Subscales: psychic (score range:0-30), neurological (score range:0-24), autonomic (score range:0-33), other (score range:0-75), global assesment by subject (score range:0-3), and global assessment by doctor (score range:0-3). Higher ratings indicate greater impairment.
Time Frame: baseline, 12 weeks
Population: All treated participants were included in the analysis population. Last observation carried forward analysis. One participant was excluded as no data for UKU were available and other participants were excluded as relevant due to absence of either baseline or post-baseline measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 151
units on a scale
  Psychic subscale, baseline; n=136 | 6.8 (4.6)
  Psychic subscale, change; n=114 | -3.5 (4.4)
  Neurological subscale, baseline; n=132 | 4.2 (2.8)
  Neurological subscale, change; n=112 | -1.2 (1.9)
  Autonomic subscale, baseline; n=132 | 1.9 (2.2)
  Autonomic subscale, change; n=113 | -0.6 (1.9)
  Other subscale, baseline; n=49 | 0.9 (2.3)
  Other subscale, baseline; n=35 | 0.2 (2.3)
  Global assessment by participant, baseline; n=150 | 0.2 (0.5)
  Global assessment by participant, change; n=129 | 0.1 (0.7)
  Global assessment by doctor, baseline; n=150 | 0.1 (0.5)
  Global assessment by doctor, change; n=129 | 0.1 (0.7)
Statistical Analysis 1: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change on the total psychic subscale score from baseline to 12-week endpoint; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for psychic subscale. A priori threshold for p-values was 0.05
Statistical Analysis 2: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change on the total neurological subscale score from baseline to 12-week endpoint; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for neurological subscale. A priori threshold for p-values was 0.05
Statistical Analysis 3: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change on the total autonomic subscale score from baseline to 12-week endpoint; Test type: Superiority or Other; p = 0.0014, t-test, 2 sided — p-value is for autonomic subscale. A priori threshold for p-values was 0.05
Statistical Analysis 4: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change on the total other subscale score from baseline to 12-week endpoint; Test type: Superiority or Other; p = 0.5586, t-test, 2 sided — p-value is for other subscale. A priori threshold for p-values was 0.05
Statistical Analysis 5: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change on the global assessment by paticipant subscale score from baseline to 12-week endpoint; Test type: Superiority or Other; p = 0.0848, t-test, 2 sided — p-value is for global assessment by paticipant. A priori threshold for p-values was 0.05
Statistical Analysis 6: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change on the global assessment by doctor subscale score from baseline to 12-week endpoint; Test type: Superiority or Other; p = 0.0263, t-test, 2 sided — p-value is for global assessment by doctor. A priori threshold for p-values was 0.05

4. Secondary Outcome: Change From Baseline on the Pittsburgh Sleep Quality Index (PSQI)
Description: Self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. 19 individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The subject self-rates each of these seven areas of sleep. Scoring of answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale. The total score is the sum of the 7 component scores (total score range: 0-21).
Time Frame: baseline, 4 weeks, 8 weeks, 12 weeks
Population: All treated participants with baseline and post-baseline data for >= 1 visit for >= 1 efficacy variable were included in the analyses (Full Analysis Set population). Last observation carried forward analysis. Excluded 2 participants (no baseline measure of PSQI) and 13 participants from calculation of change (absence of any post-baseline measure).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 149
units on a scale
  baseline, n=147 | 8.6 (3.7)
  4 weeks change, n=134 | -2.8 (3.1)
  8 weeks change, n=134 | -3.3 (3.5)
  12 weeks change, n=134 | -3.2 (3.5)
Statistical Analysis 1: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change on the Pittsburgh Sleep Quality Index from baseline to 4-week endpoint; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for 4 weeks change. A priori threshold for p-values was 0.05
Statistical Analysis 2: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change on the Pittsburgh Sleep Quality Index from baseline to 8-week endpoint; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for 8 weeks change. A priori threshold for p-values was 0.05
Statistical Analysis 3: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change on the Pittsburgh Sleep Quality Index from baseline to 12-week endpoint; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for 12 weeks change. A priori threshold for p-values was 0.05

5. Secondary Outcome: Change From Baseline to 12 Weeks on the 17-item Hamilton Depression Rating Scale (HAMD-17) Total Score
Description: The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: baseline, 12 weeks
Population: All treated participants for whom both baseline data and post-baseline data for at least 1 visit for at least one efficacy variable were available (Full analysis set population) were included in the analyses. Last observation carried forward analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 149
units on a scale
  baseline | 19.2 (3.5)
  change | -10.1 (6.5)
Statistical Analysis 1: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change on the HAMD-17 total score from baseline to 12-week endpoint; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for the HAMD-17 total score. A priori threshold for p-values was 0.05

6. Secondary Outcome: Change From Baseline to 12 Weeks on the Clinical Global Impression-Severity Scale
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: baseline, 12 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 149
units on a scale
  baseline | 4.0 (0.7)
  change | -1.5 (1.3)
Statistical Analysis 1: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change on the Clinical Global Impression-Severity scale score from baseline to end of week 12 of treatment; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for Clinical Global Impression-Severity scale - change. A priori threshold for p-values was 0.05

7. Secondary Outcome: Patient's Global Impression-Improvement at Week 12
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. Scoring: 1=very much better; 2=much better; 3=low better; 4=no change; 5=low worse; 6=much worse; 7=very much worse.
Time Frame: 12 weeks
Population: All treated participants for whom both baseline data and post-baseline data for at least 1 visit for at least one efficacy variable were available (Full analysis set population) were included in the analyses.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 149
participants
  score=1 | 5
  score=2 | 63
  score=3 | 38
  score=4 | 10
  score=5 | 3
  score=6 | 0
  score=7 | 0

8. Secondary Outcome: Change From Baseline to 12 Weeks in Beck Depression Inventory (BDI) Total Score
Description: A 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a four-point scale for each item ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: baseline, 12 weeks
Population: All treated participants for whom both baseline data and post-baseline data for at least 1 visit for at least one efficacy variable were available (Full analysis set population) were included in the analyses. Last observation carried forward analysis. 27 participants had no post baseline measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 149
units on a scale
  baseline, n=149 | 21.6 (6.1)
  change, n=122 | -12.0 (7.8)
Statistical Analysis 1: Comparison: Duloxetine; Tested was the null hypothesis that there would be no difference between baseline and post-baseline in BDI scores; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for BDI score - change. A priori threshold for p-values was 0.05

9. Secondary Outcome: Change From Baseline to 12 Weeks in Visual Analog Scale (VAS)
Description: VAS for pain consists of 6 questions that assess overall pain, headache, back pain, shoulder pain, pain interference with daily activities, and pain while awake. Participant rates pain on a 100 millimeter (mm) line between two anchors (0= no pain and 100=very severe pain). Here, the line was only 93 mm long due to an error on the clinical research form and scores were adjusted to 0 to 93.
Time Frame: baseline, 12 weeks
Population: All treated participants for whom both baseline data and post-baseline data for at least 1 visit for at least 1 efficacy variable were available (Full analysis set population) were included in the analyses. Last observation carried forward analysis. Excluded were 2 participants with only post-baseline data and 1 participant with only baseline data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 149
units on a scale
  Overall pain, baseline; n=147 | 30.5 (24.1)
  Overall pain, change; n=146 | -5.1 (20.1)
  Headaches, baseline; n=147 | 15.9 (20.3)
  Headaches, change; n=146 | -5.4 (17.1)
  Back ache, baseline; n=147 | 34.9 (27.2)
  Back ache, change; n=146 | -10.2 (20.8)
  Shoulder pain, baseline; n=147 | 26.7 (27.1)
  Shoulder pain, change; n=146 | -10.3 (22.1)
  Interference, baseline; n=147 | 30.4 (26.8)
  Interference, change; n=146 | -8.2 (22.3)
  Pain while awake, baseline; n=147 | 31.7 (25.9)
  Pain while awake, change; n=146 | -9.9 (21.8)
Statistical Analysis 1: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change from baseline to 12 weeks in VAS overall pain scores; Test type: Superiority or Other; p = 0.0027, t-test, 2 sided — p-value is for VAS overall pain score - change. A priori threshold for p-values was 0.05
Statistical Analysis 2: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change from baseline to 12 weeks in VAS headaches scores; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided — p-value is for VAS Headaches score - change. A priori threshold for p-values was 0.05
Statistical Analysis 3: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change from baseline to 12 weeks in VAS back ache scores; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for VAS back ache score - change. A priori threshold for p-values was 0.05
Statistical Analysis 4: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change from baseline to 12 weeks in VAS shoulder pain score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for VAS shoulder pain score - change. A priori threshold for p-values was 0.05
Statistical Analysis 5: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change from baseline to 12 weeks in VAS interference score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for VAS interference score - change. A priori threshold for p-values was 0.05
Statistical Analysis 6: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change from baseline to 12 weeks in VAS pain while awake score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for VAS pain while awake score - change. A priori threshold for p-values was 0.05

10. Secondary Outcome: Change From Baseline to 12 Weeks in Parkinson Disease Questionnaire - 39 Item Version (PDQ-39) Total Score
Description: The PDQ-39 has 39 items. Higher scores reflect lower quality of life. The PDQ-39 has eight subscales: mobility (10 items), activities of daily living (six items), emotional wellbeing (six items), stigma (four items), social support (three items), cognition (four items), communication (three items), and bodily discomfort (three items). Items in each subscale, as well in the total scale, can be summarized into an index and transformed linearly to a 0-100 scale.
Time Frame: baseline, 12 weeks
Population: All treated participants with both baseline data and post-baseline data for at least 1 visit for at least 1 efficacy variable were available (Full analysis set population) were included in the analyses. Last observation carried forward analysis. Excluded were 2 participants with no baseline measure and 29 participants with no post baseline measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 149
units on a scale
  baseline; n=147 | 32.9 (12.5)
  change; n=118 | -7.7 (9.9)
Statistical Analysis 1: Comparison: Duloxetine; Tested was the null hypothesis that there would be no change from baseline to 12 weeks in PDQ-39 total score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value is for PDQ-39 total score - change. A priori threshold for p-values was 0.05

11. Secondary Outcome: Average Change From Baseline to 12 Weeks in Blood Pressure
Description: For each participant, changes across individual visits were averaged to obtain 1 measurement per participant.
Time Frame: baseline through 12 weeks
Population: All treated participants were included in the analysis population. 5 participants for standing measurement and 6 participants for supine measurements were excluded from calculation of change as they had either no baseline or no post-baseline measure.
Measure: Mean (95% Confidence Interval); unit: millimeter mercury
Arm/Group | Duloxetine
Number analyzed (Participants) | 151
millimeter mercury
  systolic blood pressure, standing; n=146 | -0.17 (8.03) [-1.49 to 1.14]
  diastolic blood pressure, standing; n=146 | 0.12 (6.16) [-0.89 to 1.13]
  systolic blood pressure, supine; n=145 | -0.30 (8.71) [-1.73 to 1.13]
  diastolic blood pressure, supine; n=145 | -0.45 (6.29) [-1.48 to 0.58]

12. Secondary Outcome: Average Change From Baseline to 12 Weeks in Heart Rate
Description: For each participant, changes across individual visits were averaged to obtain 1 measurement per participant.
Time Frame: baseline through 12 weeks
Population: All treated participants were included in the analysis population. 6 participants were excluded from calculation of change as they had either no baseline or post-baseline measure.
Measure: Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | Duloxetine
Number analyzed (Participants) | 151
beats per minute
  standing, n=145 | 1.61 (7.7) [0.71 to 2.51]
  supine, n=145 | 1.16 (7.9) [0.35 to 1.97]

13. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms (ECG) During the 12 Week Study
Description: Included were participants with normal ECG at baseline who developed abnormal ECGs during the study.
Time Frame: baseline through 12 weeks
Population: All treated participants were included in the analysis population. 54 participants were excluded from calculation of change as they had abnormal ECG at baseline, no baseline measure, or no post-baseline measure.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 151
participants | 3

14. Secondary Outcome: Laboratory Analytes
Description: Laboratory analytes were collected to assess adverse events which are listed in the reported adverse events section.
Time Frame: baseline through 12 weeks
Population: All enrolled participants for whom both baseline data and post-baseline data were available were included in the analyses.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants Who Responded to Treatment by 12 Weeks
Description: Response was defined as a >= 50% reduction in 17-item Hamilton Depression rating scale (HAMD) scores. The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: 12 weeks
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 149
participants | 90

16. Secondary Outcome: Number of Participants Who Reached Remission by 12 Weeks
Description: Remission was defined as reaching a 17-item Hamilton Depression Rating Scale (HAMD) total score <=7. The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: 12 weeks
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 149
participants | 68

ADVERSE EVENTS:
Arm/Group | Duloxetine
Serious Adverse Events (participants affected / at risk) | 3/151
Other Adverse Events (participants affected / at risk) | 39/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=151)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) — This event resulted in death.
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) — This event resulted in death after completing the 12 week study period but within 30 days after completing the study.
Renal failure acute (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=151)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Aptyalism (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6)
Asthenia (General disorders) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Somnolence (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Psychotic disorder (Psychiatric disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days